CLINICAL TRIAL: NCT00736944
Title: Trial to Determine the CR Rate at the Primary Tumor Site After 2 Cycles of Induction Chemo With Abraxane, Cetuximab, Cisplatin, & 5-FU for Advanced Head & Neck Carcinoma Treated With Definitive Concurrent Cisplatin & Radiation Therapy
Brief Title: Trial of 2 Cycles of Induction Chemo With Abraxane, Cetuximab, Cisplatin, & 5-FU for Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-0911 / 201105501
Record Dates: First submitted 2008-08-13; First posted 2008-08-18 (Estimated); Results first posted 2014-01-07 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Albumin-Bound Paclitaxel; Cetuximab; Cisplatin; Fluorouracil; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Induction chemotherapy followed by Radiation therapy plus Cisplatin
  Induction chemotherapy:
  Abraxane 100 mg/m2 IVPB, Day 1, 8, and 15 of cycles 1, 2, and 3. Cetuximab 400 mg/m2 IVPB, Day 1, cycle 1. Cetuximab 250 mg/m2 IVPB, Day 8 and 15 cycle 1, 2 and 3. Cisplatin 75 mg/m2 IVPB, Day 1, cycles 1, 2, and 3. 5-FU 750 mg/m2 CIVI, Day 1, 2 and 3, cycles 1, 2, and 3.
  Post-Induction:
  Radiation - Monday-Friday weeks 1-7 with concurrent Cisplatin 100 mg/m2 IVPB on radiation day 1, 22, and 42.
  Interventions: Drug: Abraxane; Drug: Cetuximab; Drug: Cisplatin; Drug: 5-FU; Radiation: Radiation (Post induction)
- 2 (Experimental): Induction chemotherapy followed by Radiation therapy plus Cetuximab
  Induction chemotherapy:
  Abraxane 100 mg/m2 IVPB, Day 1, 8, and 15 of cycles 1, 2, and 3. Cetuximab 400 mg/m2 IVPB, Day 1, cycle 1. Cetuximab 250 mg/m2 IVPB, Day 8 and 15 cycle 1, 2 and 3. Cisplatin 75 mg/m2 IVPB, Day 1, cycles 1, 2, and 3. 5-FU 750 mg/m2 CIVI, Day 1, 2 and 3, cycles 1, 2, and 3.
  Post-Induction:
  Radiation - Monday-Friday weeks 1-7 with concurrent Cetuximab (for patients who cannot receive cisplatin) will begin (+/- 3 days) before starting radiation therapy at 400 mg/m2 IVPB. Subsequent doses of cetuximab will be given weekly at 250 mg/m2 IVPB
  Interventions: Drug: Abraxane; Drug: Cetuximab; Drug: Cisplatin; Drug: 5-FU; Radiation: Radiation (Post induction)

INTERVENTIONS:
Drug: Abraxane — 100 mg/m2 IVPB, Day 1, 8 and 15 of cycles 1, 2, and 3
Drug: Cetuximab — 400 mg/m2 IVPB, Day 1, cycle 1
Drug: Cetuximab — 250 mg IVPB, Day 8 and 15 cycle 1, Day 1, 8 and 15 of cycles 2 and 3
Drug: Cisplatin — 75 mg/m2 IVPB Day 1, cycles 1, 2 and 3
Drug: 5-FU — 750 mg/m2 CIVI Day 1, 2 and 3, cycles 1, 2 and 3
Radiation: Radiation (Post induction) — Monday-Friday, weeks 1-7
Drug: Cisplatin — (Post induction) Cisplatin 100 mg/m2 IVPB on radiation day 1, 22 and 42
  Arms: 1
Drug: Cetuximab — (Post-induction) Cetuximab (for patients who cannot receive cisplatin) will begin (+/- 3 days) before starting radiation therapy at 400 mg/m2 IVPB. Subsequent doses of cetuximab will be given weekly at 250 mg/m2 IVPB
  Arms: 2

SUMMARY:
This phase two trial will determine the tumor response rate at the primary site and at involved regional nodes to two cycles of an IC regimen of weekly Abraxane and cetuximab given in combination with cisplatin and 5-FU in patients with local regionally advanced HNSCC.

DETAILED DESCRIPTION:
Primary objective:

To determine the clinical CR rate (CR-p) at the primary tumor site to an IC regimen of weekly Abraxane and cetuximab with CF (ACCF) given for two cycles (over 6 weeks) in patients with locally advanced non-metastatic HNSCC. The assessment of primary tumor site response will be performed by the treating physician by careful clinical examination using WHO criteria. Radiographic studies will also be performed to assess primary tumor site response but will be used primarily to confirm lack of disease progression that may not be detected based on clinical examination alone.

The secondary objectives include:

* Document the clinical PR rate (PR-p) at the primary tumor site with this IC regimen
* Document the clinical CR and PR rates at the involved regional nodes (CR-n and PR-n) with this IC regimen
* Document the clinical overall CR rate (CR-o) (defined as achievement of a CR at the primary tumor site and at the involved regional nodes) and the clinical overall PR rate (PR-o) with this IC regimen
* Document the CR (CR-p, CR-n, and CR-o) and PR (PR-p, PR-n, and PR-o) rates by FDG uptake on PET scan after this IC regimen
* Document radiographic CR (CR-p, CR-n, and CR-o) and PR (PR-p, PR-n, and PR-o) rates as assessed by conventional CT scan using RECIST criteria after this IC regimen.
* Correlate primary tumor site, nodal and overall tumor response rates based on WHO criteria of assessment with that based on CT scan and FDG-PET/CT.
* Document and quantify SPARC expression by IHC in primary tumor tissue obtained at baseline in each patient and attempt to correlate these results with primary tumor site response to ACCF.
* Document and grade AE's with this IC regimen with a pre-planned safety analysis after the first ten patients have completed the IC regimen.
* Determine the overall survival (OS), disease-free survival (DFS), and progression-free survival (PFS) of this patient population.

ELIGIBILITY:
Inclusion

* Selected Stages 3 and 4a/b HNSCC: All patients must have T2-T4 primary tumors. Patients with T1 tumors will be excluded. Although most of these patients will have regional nodal disease, patients with no nodal disease will also be eligible.
* Oropharynx, hypopharynx, larynx, and oral cavity sub-sites only. Patients with nasopharyngeal, sinus and other sub-sites of the head and neck, or unknown primary SCC of the head and neck will NOT be eligible.
* Age ≥18 years
* Signed informed consent.
* ECOG Performance Status (PS) of 0-2 (Appendix 1).
* Adequate vital organ function (serum creatinine < 1.8 mg/dl, total bilirubin </= 1.5 mg/dl, ALT and AST </= 2.5 x ULN, alkaline phosphatase </= 2.5 x ULN) and hematopoietic function (ANC >/= 1500/ul, Platelets > 100,000/ul, HGB > 9.0 g/dl).
* Patients with reproductive potential must use an effective method of contraception to avoid pregnancy for the duration of the trial and for three months after completing treatment.
* If female of childbearing potential, the patient must have a negative pregnancy test.

Exclusion Criteria:

* Peripheral neuropathy > Grade 1.
* Prior chemotherapy, EGFR targeted therapy or radiation therapy for HNSCC.
* History of prior invasive malignancy diagnosed within the last three years other than local stage non-melanoma skin cancer.
* Be taking cimetidine or allopurinol. Patients must discontinue taking the medication for one week before receiving treatment with Abraxane.
* Be taking cimetidine or allopurinol. Patients must discontinue taking the medication for one week before receiving treatment with Abraxane.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-12-19 (Actual); Primary Completion 2010-08-31 (Actual); Study Completion 2020-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Adkins, M.D., Principal Investigator — Washington Univerisity
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Department of Veterans Affairs Laryngeal Cancer Study Group; Wolf GT, Fisher SG, Hong WK, Hillman R, Spaulding M, Laramore GE, Endicott JW, McClatchey K, Henderson WG. Induction chemotherapy plus radiation compared with surgery plus radiation in patients with advanced laryngeal cancer. N Engl J Med. 1991 Jun 13;324(24):1685-90. doi: 10.1056/NEJM199106133242402. PMID 2034244
- [Background] JCO 12:1592, 1194
- [Background] Hitt R, Lopez-Pousa A, Martinez-Trufero J, Escrig V, Carles J, Rizo A, Isla D, Vega ME, Marti JL, Lobo F, Pastor P, Valenti V, Belon J, Sanchez MA, Chaib C, Pallares C, Anton A, Cervantes A, Paz-Ares L, Cortes-Funes H. Phase III study comparing cisplatin plus fluorouracil to paclitaxel, cisplatin, and fluorouracil induction chemotherapy followed by chemoradiotherapy in locally advanced head and neck cancer. J Clin Oncol. 2005 Dec 1;23(34):8636-45. doi: 10.1200/JCO.2004.00.1990. Epub 2005 Nov 7. PMID 16275937
- [Background] Burtness B, Goldwasser MA, Flood W, Mattar B, Forastiere AA; Eastern Cooperative Oncology Group. Phase III randomized trial of cisplatin plus placebo compared with cisplatin plus cetuximab in metastatic/recurrent head and neck cancer: an Eastern Cooperative Oncology Group study. J Clin Oncol. 2005 Dec 1;23(34):8646-54. doi: 10.1200/JCO.2005.02.4646. PMID 16314626
- [Background] Kuperman, et al ASCO 2007
- [Background] Kies, et al ASCO 2006
- [Background] ten Tije AJ, Verweij J, Loos WJ, Sparreboom A. Pharmacological effects of formulation vehicles : implications for cancer chemotherapy. Clin Pharmacokinet. 2003;42(7):665-85. doi: 10.2165/00003088-200342070-00005. PMID 12844327
- [Background] Sparreboom A, van Zuylen L, Brouwer E, Loos WJ, de Bruijn P, Gelderblom H, Pillay M, Nooter K, Stoter G, Verweij J. Cremophor EL-mediated alteration of paclitaxel distribution in human blood: clinical pharmacokinetic implications. Cancer Res. 1999 Apr 1;59(7):1454-7. PMID 10197613
- [Background] Winer EP, Berry DA, Woolf S, Duggan D, Kornblith A, Harris LN, Michaelson RA, Kirshner JA, Fleming GF, Perry MC, Graham ML, Sharp SA, Keresztes R, Henderson IC, Hudis C, Muss H, Norton L. Failure of higher-dose paclitaxel to improve outcome in patients with metastatic breast cancer: cancer and leukemia group B trial 9342. J Clin Oncol. 2004 Jun 1;22(11):2061-8. doi: 10.1200/JCO.2004.08.048. PMID 15169793
- [Background] van Tellingen O, Huizing MT, Panday VR, Schellens JH, Nooijen WJ, Beijnen JH. Cremophor EL causes (pseudo-) non-linear pharmacokinetics of paclitaxel in patients. Br J Cancer. 1999 Sep;81(2):330-5. doi: 10.1038/sj.bjc.6690696. PMID 10496361
- [Background] Desai N, et al SABCS Dec, 2003
- [Background] Gradishar WJ, Tjulandin S, Davidson N, Shaw H, Desai N, Bhar P, Hawkins M, O'Shaughnessy J. Phase III trial of nanoparticle albumin-bound paclitaxel compared with polyethylated castor oil-based paclitaxel in women with breast cancer. J Clin Oncol. 2005 Nov 1;23(31):7794-803. doi: 10.1200/JCO.2005.04.937. Epub 2005 Sep 19. PMID 16172456
- [Background] Gradishar,et al SABCS 2006
- [Background] SABCS 2006
- [Background] Kato Y, Nagashima Y, Baba Y, Kawano T, Furukawa M, Kubota A, Yanoma S, Imagawa-Ishiguro Y, Satake K, Taguchi T, Hata R, Mochimatsu I, Aoki I, Kameda Y, Inayama Y, Tsukuda M. Expression of SPARC in tongue carcinoma of stage II is associated with poor prognosis: an immunohistochemical study of 86 cases. Int J Mol Med. 2005 Aug;16(2):263-8. PMID 16012759
- [Background] Mendez E, et al Cancer 95:1482-1494, 2005
- [Background] Desai N, et al SABCS Dec, 2004
- [Derived] Adkins D, Ley J, Oppelt P, Wildes TM, Gay HA, Daly M, Rich J, Paniello RC, Jackson R, Pipkorn P, Nussenbaum B, Trinkaus K, Thorstad W. nab-Paclitaxel-based induction chemotherapy with or without cetuximab for locally advanced head and neck squamous cell carcinoma. Oral Oncol. 2017 Sep;72:26-31. doi: 10.1016/j.oraloncology.2017.07.001. Epub 2017 Jul 8. PMID 28797458
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was open from 12/19/08-10/18/11 at the Siteman Cancer Center (a medical clinic).
Groups:
- Induction Chemo + RT + Cisplatin or Cetuximab: Induction chemotherapy:
  Abraxane 100 mg/m2 IVPB, Day 1, 8, and 15 of cycles 1, 2, and 3. Cetuximab 400 mg/m2 IVPB, Day 1, cycle 1. Cetuximab 250 mg/m2 IVPB, Day 8 and 15 cycle 1, 2 and 3. Cisplatin 75 mg/m2 IVPB, Day 1, cycles 1, 2, and 3. 5-FU 750 mg/m2 CIVI, Day 1, 2 and 3, cycles 1, 2, and 3.
  Post-Induction:
  Radiation - Monday-Friday weeks 1-7 with concurrent Cisplatin 100 mg/m2 IVPB on radiation day 1, 22, and 42 or Cetuximab 250 mg/m2 IVPB weekly Q8W.
Period: Induction
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Started | 30
Completed | 29
Not Completed | 1
Not completed — Death | 1
Period: Definitive Treatment
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Started | 29
Completed | 28
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 54.5 [39 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Clinical Complete Response Rate at the Primary Tumor
Description: Clinical exam included laryngoscopy in office or operating room.
  Complete response rate includes complete response (CR) which is defined as 100% decrease in tumor size and it also includes near complete response (near CR) defined as 95-99% decrease in tumor size.
Time Frame: post-2 cycles of induction (approximately 42 days from start of treatment)
Population: All patients who completed 2 cycles of induction therapy.
Measure: Number; unit: participants
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 30
participants | 16

2. Secondary Outcome: Clinical Partial Response Rate at the Primary Tumor
Description: Clinical exam included laryngoscopy in office or operating room.
  Partial response rate (PR) defined as 50% to 94% decrease in tumor size.
Time Frame: post-2 cycles of induction therapy (approximately 42 days from start of treatment)
Population: Participants who completed 2 cycles of induction therapy
Measure: Number; unit: participants
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 30
participants | 14

3. Secondary Outcome: Clinical Complete and Partial Response Rates to the Involved Regional Nodes
Description: Clinical exam consisted of physical exam of neck in office.
  Complete response rate includes complete response (CR) which is defined as 100% decrease in tumor size and near complete response (near CR) defined as 95-99% decrease in tumor size.
  Partial response rate defined as 50% to 94% decrease in tumor size.
Time Frame: post-2 cycles of induction therapy (approximately 42 days from start of treatment)
Population: Twelve patients were not evaluable because of initial absence of nodal disease on clinical exam.
Measure: Number; unit: participants
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 18
participants
  Complete response | 11
  Partial response | 7

4. Secondary Outcome: Clinical Overall Complete and Partial Response Rates
Description: Clinical exam included laryngoscopy in office or operating room.
  Clinical exam consisted of physical exam of neck in office.
  Complete response rate includes complete response (CR) which is defined as 100% decrease in tumor size and it also includes near complete response (near CR) defined as 95-99% decrease in tumor size.
  Partial response rate defined as 50% to 94% decrease in tumor size.
Time Frame: post-2 cycles of induction therapy (approximately 42 days)
Measure: Number; unit: participants
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 30
participants
  Overall complete response | 13
  Overall partial response | 17

5. Secondary Outcome: Complete and Partial Response Rates of Primary Tumor by FDG Uptake on PET Scan
Description: Complete response rate defined as complete resolution of the metabolically active primary tumor.
  Partial response rate defined as 20% or greater decrease in maximum SUV [SUV g/ml) = ROI activity (mCi/ml) / (injected dose (mCi/body weight(g))] from baseline. No unequivocal metabolic progression of non-target disease, and no unequivocal new lesions.
Time Frame: post-2 cycles of induction therapy (approximately 42 days from start of treatment)
Population: Two patients were not evaluable for this outcome. One patient's insurance company denied coverage for the PET scan so the PET scan was not performed. The other patient only had neck nodes that were clearly measurable on the PET scan, the primary site could not be measured on the PET scan.
Measure: Number; unit: participants
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 28
participants
  Complete response | 9
  Partial response | 17

6. Secondary Outcome: Complete and Partial Response Rates of Involved Lymph Nodes by FDG Uptake on PET Scan
Description: as for outcome 5
Time Frame: post-2 cycles of induction therapy (approximately 42 days from start of treatment)
Population: Five patients were not evaluable for this outcome because these patients did not have any involved lymph nodes that could be measured.
Measure: Number; unit: participants
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 25
participants
  Complete response | 9
  Partial response | 14

7. Secondary Outcome: Radiographic Complete and Partial Response Rates of Primary Tumor as Assessed by Conventional CT Scan Using RECIST Criteria
Description: Complete response rate per RECIST criteria is defined as disappearance of all target lesions.
  Partial response rate per RECIST criteria is defined as at least a 30% decrease in the sum of the longest diameter of target lesions taking as reference the baseline sum longest diameter.
Time Frame: post-2 cycles of induction therapy (approximately 42 days from start of treatment)
Population: Two patients were not evaluable for this outcome. The first patient didn't have primary site disease that could be measured by RECIST. The second patient had primary site disease but it could not be clearly measured by CT. This disease was noted as a non-target lesion as present at baseline.
Measure: Number; unit: participants
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 28
participants
  Complete response | 10
  Partial response | 11

8. Secondary Outcome: Radiographic Complete and Partial Response Rates of Involved Lymph Nodes as Assessed by Conventional CT Scan Using RECIST Criteria
Description: as for outcome 7
Time Frame: post-2 cycles of induction therapy (approximately 42 days from start of treatment)
Population: Six patients were not evaluable for this outcome. Five of these patients did not have any involved lymph nodes available to evaluate. The sixth patient did not have involved lymph nodes that were clearly measurable by CT and RECIST.
Measure: Number; unit: participants
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 24
participants
  Complete response | 7
  Partial response | 12

9. Secondary Outcome: Radiographic Overall Complete and Partial Response Rates as Assessed by Conventional CT Scan Using RECIST Criteria
Description: as for outcome 7
Time Frame: post-2 cycles of induction therapy (approximately 42 days from start of treatment)
Population: One patient was not evaluable for this outcome. This patient had primary site disease that could not be clearly measured per CT and was listed as a non-target lesion.
Measure: Number; unit: participants
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 29
participants
  Overall complete response | 4
  Overall partial response | 14

10. Secondary Outcome: Correlate Primary Tumor Site Response Rates Based on Visual Categorical Criteria of Assessment With That Based on CT Scan and FDG-PET/CT
Description: In the future, primary tumor site, nodal, and OTR by VCR (CR-x or PR-x = Y or N) will be compared with response based on CT scan (CR-x or PR-x = Y or N) using a test for difference in paired, binary values. Median standardized uptake value of FDG measured by PET/CT will be compared among those with or without response (CR-x or PR-x) using nonparametric Wilcoxon-Mann-Whitney tests.
  We are releasing results based on comparing actual responses from visual categorical response, CT scan, and FDG-PET/CT scan after 2 cycles.
Time Frame: post-2 cycles of induction therapy (approximately 42 days from start of treatment)
Population: 2 patients were not evaluable for the CT Scan of this outcome because they did not have primary disease that could be measured per RECIST. 2 patients were not evaluable for PET scan of this outcome because one patient's insurance company denied coverage and the other patient did not have primary site disease.
Measure: Number; unit: percentage of participants
Arm/Group | Clinical Examination | CT Scan | FDG-PET/CT
Number analyzed (Participants) | 30 | 28 | 28
percentage of participants
  Complete Response | 53 | 33 | 32
  Partial Response | 47 | 41 | 61
  Stable Disease/Progressive Disease | 0 | 26 | 7

11. Secondary Outcome: Correlate Nodal Response Rates Based on Visual Categorical Criteria of Assessment With That Based on CT Scan and FDG-PET/CT
Description: In the future, primary tumor site, nodal, and overall tumor response by visual categorical response (CR-x or PR-x = yes or no) will be compared with response based on CT scan (CR-x or PR-x = yes or no) using a test for difference in paired, binary values (e.g., McNemar's test). Median standardized uptake value of FDG measured by PET/CT will be compared among those with or without response (CR-x or PR-x) using nonparametric Wilcoxon-Mann-Whitney tests. At this point, we are releasing results based on comparing actual responses from visual categorical response, CT scan, and FDG-PET/CT scan after 2 cycles of induction.
Time Frame: post-2 cycles of induction therapy (approximately 42 days from start of treatment)
Population: 12 patients were not evaluable for VSR because they did not have nodal disease. 6 patients were not evaluable for CT scan because 5 patients did not have nodal disease and 1 patient didn't have measurable nodal disease. 5 patients were not evaluable for PET because 5 patients did not have nodal disease.
Measure: Number; unit: percentage of participants
Arm/Group | Clinical Examination | CT Scan | FDG-PET/CT
Number analyzed (Participants) | 18 | 24 | 25
percentage of participants
  Complete Response | 61 | 30 | 36
  Partial Response | 39 | 48 | 56
  Stable Disease/Progressive Disease | 0 | 22 | 8

12. Secondary Outcome: Correlate Overall Tumor Response Rates Based on Visual Categorical Criteria of Assessment With That Based on CT Scan and FDG-PET/CT
Description: as for outcome 11
Time Frame: post-2 cycles of induction therapy (approximately 42 days from start of treatment)
Population: 1 patient was not evaluable for CT scan because the primary site could not be clearly measured and was noted as non-target lesion. 1 patient was not evaluable for PET scan because the patient's insurance company denied coverage.
Measure: Number; unit: percentage of participants
Arm/Group | Clinical Examination | CT Scan | FDG-PET/CT
Number analyzed (Participants) | 30 | 29 | 29
percentage of participants
  Complete Response | 43 | 14 | 24
  Partial Response | 57 | 50 | 66
  Stable Disease/Progressive Disease | 0 | 36 | 10

13. Secondary Outcome: Correlate SPARC Expression by Immunohistochemistry (IHC) in Baseline Primary Tumor Tissue With Primary Tumor Site Complete Response Rate to Induction Chemotherapy
Description: SPARC expression = Proportion of tumor cells SPARC-positive in 10 high-power fields
Time Frame: post-2 cycles of induction therapy (approximately 42 days from start of treatment)
Population: Patients who had available tumor tissue for SPARC testing and were complete responders.
Measure: Number; unit: participants
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 15
participants
  Negative staining | 14
  1+ staining (0%-24%) | 0
  2+ staining (25%-49%) | 1
  3+ staining (50%-74%) | 0
  4+ staining (75%-100%) | 0

14. Secondary Outcome: Correlate SPARC Expression by Immunohistochemistry (IHC) in Baseline Primary Tumor Tissue With Primary Tumor Site Partial Response Rate to Induction Chemotherapy
Description: SPARC expression = Proportion of tumor cells SPARC-positive in 10 high-power fields
Time Frame: post-2 cycles of induction therapy (approximately 42 days from start of treatment)
Population: Patients who had available tumor tissue for SPARC testing and were partial responders.
Measure: Number; unit: participants
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 13
participants
  Negative staining | 6
  1+ staining (0%-24%) | 4
  2+ staining (25%-49%) | 1
  3+ staining (50%-74%) | 2
  4+ staining (75%-100%) | 0

15. Secondary Outcome: Correlate SPARC Expression (Intensity of Staining) by Immunohistochemistry (IHC) in Baseline Primary Tumor Tissue With Primary Tumor Site Complete Response Rate to Induction Chemotherapy
Description: SPARC expression = intensity of SPARC staining in tumor
Time Frame: post-2 cycles of induction therapy (approximately 42 days from start of treatment)
Population: Patients who had available tumor tissue for SPARC testing and were complete responders.
Measure: Number; unit: participants
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 15
participants
  Negative staining | 14
  1+ staining (weak) | 0
  2+ staining (moderate) | 1
  3+ staining (strong) | 0

16. Secondary Outcome: Correlate SPARC Expression (Intensity of Staining) by Immunohistochemistry (IHC) in Baseline Primary Tumor Tissue With Primary Tumor Site Partial Response Rate to Induction Chemotherapy
Description: SPARC expression = intensity of SPARC staining in tumor
Time Frame: post-2 cycles of induction therapy (approximately 42 days from start of treatment)
Population: Patients who had available tumor tissue for SPARC testing and were partial responders.
Measure: Number; unit: participants
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 13
participants
  Negative staining | 6
  1+ staining (weak) | 2
  2+ staining (moderate) | 4
  3+ staining (strong) | 1

17. Secondary Outcome: Adverse Events Experienced During Induction Chemotherapy in the First Ten Patients for a Pre-planned Safety Analysis
Time Frame: completion of the first 10 patients induction chemotherapy
Measure: Number; unit: participants
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 10
participants
  Allergic reaction/hypersensitivity | 1
  Other allergic reaction:cipro | 1
  Other allergic reaction:hives | 1
  Hypotension | 1
  INR | 1
  Fatigue | 10
  Alopecia | 5
  Chelitis | 1
  Dry skin | 1
  Rash | 1
  Rash:acneiform | 7
  Rash:penile (unconfirmed HSV) | 1
  Anorexia | 1
  Colitis | 2
  Constipation | 1
  Dehydration | 1
  Dental:teeth | 1
  Diarrhea | 1
  Hemorrhoids | 1
  Nausea | 9
  Taste alteration | 1
  Vomiting | 1
  Other:soft stools | 1
  Hemoglobin | 8
  Leukocytes (WBC) | 8
  Lymphopenia | 8
  Neutrophils (ANC) | 8
  Platelets | 2
  Hemmorrhage:nose | 1
  Alkaline phosphatase | 3
  SGPT (ALT) | 2
  Infection other:sinus infection | 1
  Edema:limb | 2
  Albumin, low | 1
  Calcium, low | 5
  Magnesium, low | 4
  Potassium, low | 3
  Potassium, high | 2
  Sodium, low | 3
  Phosphorus | 1
  Dizziness | 1
  Mood alteration:anger | 1
  Neuropathy:sensory (peripheral) | 1
  Vision-photophobia | 1
  Pain:thigh | 1
  Pain:tumor pain | 1
  Hiccoughs (hiccups) | 1
  Obstruction/stenosis of airway:trachea | 2
  Creatinine | 4
  GFR | 2
  Renal failure | 1
  Thrombosis/thrombus/embolism | 1

18. Secondary Outcome: Overall Survival
Description: Time from diagnosis to death or to last follow-up alive.
Time Frame: 10 years from completion of treatment
Measure: Mean (Standard Error); unit: months
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 30
months | 83.960 (5.384)

19. Secondary Outcome: Disease Free Survival
Description: Time from complete response to death from any cause, to disease progression or to last follow-up alive.
Time Frame: 10 years from completion of treatment
Measure: Mean (Standard Error); unit: months
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 30
months | 93.529 (3.462)

20. Secondary Outcome: Time to Progression
Description: Time from initiation of induction chemotherapy to death due to disease progression, to disease progression, or to last follow-up alive.
Time Frame: 10 years from completion of treatment
Measure: Mean (Standard Error); unit: months
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 30
months | 38.675 (1.485)

21. Other Pre Specified Outcome: Overall Complete and Partial Response Rates by FDG Uptake on PET Scan
Description: as for outcome 5
Time Frame: post-2 cycles of induction therapy (approximately 42 days from start of treatment)
Population: One patient was not evaluable for this outcome. This patient's insurance company denied coverage for the post-cycle 2 timepoint and because of this was not included in this overall response rate for PET scan.
Measure: Number; unit: participants
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Number analyzed (Participants) | 29
participants
  Overall complete response | 7
  Overall partial response | 19

ADVERSE EVENTS:
Time Frame: From time of consent through completion of induction chemotherapy.
Description: Serious adverse events are events grade 3 or higher.
  Lab results, treatment records, and dictations reviewed weekly.
Arm/Group | Induction Chemo + RT + Cisplatin or Cetuximab
Serious Adverse Events (participants affected / at risk) | 19/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Chemo + RT + Cisplatin or Cetuximab (N=30)
Allergic reaction/hypersensitivity (Immune system disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Leukocytes (WBC) (Investigations) | 3 (3)
Lymphopenia (Investigations) | 4 (4)
Neutrophils (ANC) (Investigations) | 5 (5)
Calcium, low (Metabolism and nutrition disorders) | 2 (2)
Potassium, low (Metabolism and nutrition disorders) | 3 (3)
Sodium, low (Metabolism and nutrition disorders) | 1 (1)
Phosphorus, low (Metabolism and nutrition disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Supraventricular and nodal arrhythmia: atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac ischemia (Cardiac disorders) | 1 (1)
Rash: acneiform (Skin and subcutaneous tissue disorders) | 4 (4)
Mucositis (Gastrointestinal disorders) | 1 (1)
Platelets (Investigations) | 1 (1)
Infection with normal ANC-rectal abscess (Infections and infestations) | 1 (1)
Infection with grade 4 neutrophils:lung-pneumonia (Infections and infestations) | 1 (1)
Albumin, low (Metabolism and nutrition disorders) | 1 (1)
Glucose, high (Metabolism and nutrition disorders) | 1 (1)
Cerebrovascular ischemia (Nervous system disorders) | 1 (1)
Pain:chest (Cardiac disorders) | 1 (1)
Thrombosis/thrombus/embolism-vascular access device (Vascular disorders) | 4 (4)
Hemoglobin (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Chemo + RT + Cisplatin or Cetuximab (N=30)
Allergic reaction/hypersensitivity (Immune system disorders) | 2 (2)
INR (Investigations) | 3 (3)
PTT (Investigations) | 2 (2)
Fatigue (General disorders) | 19 (19)
Weight loss (Investigations) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11)
Rash:acneiform (Skin and subcutaneous tissue disorders) | 20 (20)
Rash:penile (unconfirmed HSV) (Skin and subcutaneous tissue disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 7 (7)
Dental:teeth (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 13 (13)
Heartburn (Gastrointestinal disorders) | 3 (3)
Mucositis (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 19 (19)
Vomiting (Gastrointestinal disorders) | 5 (5)
Hemoglobin (Investigations) | 26 (26)
Leukocytes (WBC) (Investigations) | 21 (21)
Lymphopenia (Investigations) | 16 (16)
Neutrophils (ANC) (Investigations) | 15 (15)
Platelets (Investigations) | 8 (8)
Hemorrhage:nose (Blood and lymphatic system disorders) | 3 (3)
Alkaline phosphatase (Investigations) | 6 (6)
SGOT (AST) (Investigations) | 3 (3)
SGPT (ALT) (Investigations) | 10 (10)
Edema:limb (General disorders) | 3 (3)
Albumin, low (Metabolism and nutrition disorders) | 6 (6)
Calcium, low (Metabolism and nutrition disorders) | 11 (11)
Glucose, high (Metabolism and nutrition disorders) | 5 (5)
Magnesium, low (Investigations) | 9 (9)
Potassium, low (Investigations) | 5 (5)
Potassium, high (Investigations) | 3 (3)
Sodium, low (Investigations) | 6 (6)
Dizziness (Nervous system disorders) | 3 (3)
Neuropathy:sensory (peripheral) (Nervous system disorders) | 6 (6)
Pain:tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccoughs (hiccups) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine (Investigations) | 7 (7)
GFR (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No